CLINICAL TRIAL: NCT02958878
Title: Preoperative Administration of Tamsulosin for Prevention of Post Operative Urinary Retention in Males Undergoing Elective Inguinal Hernia Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ascension Health (Industry)
Responsible Party: Principal Investigator, Anthony Tabatabai, General Surgery Resident, Ascension Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GenesysRMC
Record Dates: First submitted 2016-11-05; First posted 2016-11-08 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Postoperative Urinary Retention
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Tamsulosin 0.4mg given the night before surgery and another dose the day of surgery in the morning.
  Interventions: Drug: Tamsulosin
- B (Placebo Comparator): Placebo medication given the night before surgery and another dose the day of surgery in the morning
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Tamsulosin
  Other Names: Flomax
  Arms: A
Drug: Placebo Oral Capsule
  Arms: B

SUMMARY:
Double blinded, randomized controlled prospective study looking at 2 preoperative doses of Tamsulosin an alpha-adrenergic blocker in preventing post-operative urinary retention. A previous study was conducted called "Effectiveness of tamsulosin inprevention of postoperative urinary retention: a randomized double-blind-placebo controlled study" This study involved a tertiary care center involving mostly urological surgical procedures. We look to specifically look at inguinal hernia surgeries in males. The aim of this study is to compare the prophylactic effect of tamsulosin with placebo on postoperative urinary retention. The drug is FDA approved for benign prostatic hypertrophy and urinary retention. It is on formulary at Genesys. Currently there is no standard procedure of prophylactic tamsulosin for urinary retention. Most often post operative patients are given tamsulosin to augment smooth muscle relaxation and spontaneous voiding if the patient is having urinary retention post operatively. We often straight catheterize patients once and start tamsulosin with the goal of avoiding urinary retention and future straight catheterizations or placement of foley catheters

ELIGIBILITY:
Inclusion Criteria:

* healthy males, who are not taking Tamsulosin regularly who are undergoing elective inguinal hernia repair (laparoscopic, open, and robotic assisted)

Exclusion Criteria:

* Patients who are already taking tamsulosin, terazosin (alpha blocker treatement for BPH) , finasteride, dutasteride ( both 5 alpha reductase inhibitors), sulfa allergy, and lactose allergy

Min Age: 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
number of Urinary Retention | within 72 hours of surgery
  If patients have urinary retention post operatively

SECONDARY OUTCOMES:
placebo vs tamsulosin | within 72 hours of surgery

IPD SHARING:
Plan to Share IPD: No